CLINICAL TRIAL: NCT03664050
Title: Laparoscopic Ovarian Drilling Versus Letrozole In Clomiphene Citrate Resistant Polycystic Ovary: A Randomized Controlled Trial
Brief Title: Laparoscopic Ovarian Drilling Versus Letrozole In Clomiphene Citrate Resistant Polycystic Ovary
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Shafy El Shahawy, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOD
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Induction of Ovulation
Keywords: letrozol; laparoscopic ovarian drilling
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A Letrozole group (Experimental): 2.5 mg letrozole oral tablets will be administered on the 2nd -3rd day of menses and then every day for 5 days.
  Interventions: Drug: group A 2.5 mg letrozole oral tablets
- Group B laparoscopic ovarian drilling group (Active Comparator): bilateral laparoscopic ovarian drilling, each ovary will be cauterized at 4 points, each for 4 sec at 40 W, at a depth of 7-8 mm and a diameter of 3-5 mm, using a monopolar electrosurgical needle according to the size of each ovary.
  Interventions: Procedure: laparoscopic ovarian drilling

INTERVENTIONS:
Drug: group A 2.5 mg letrozole oral tablets — 2.5 mg letrozole oral tablets will be administered on the 2nd-3rd day of menses and then every day for 5 days. Treatment will be repeated for up to three cycles if the patient failed to conceive.
  Arms: Group A Letrozole group
Procedure: laparoscopic ovarian drilling — Bilateral laparoscopic ovarian drilling, each ovary will be cauterized at 4 points, each for 4 sec at 40 W, at a depth of 7-8 mm and a diameter of 3-5 mm, using a monopolar electrosurgical needle according to the size of each ovary.
  Arms: Group B laparoscopic ovarian drilling group

SUMMARY:
The aim of this work is to compare the clinical outcomes of letrozole with laparoscopic ovarian drilling (LOD) in patients with clomiphene-citrate-resistant polycystic ovary syndrome (PCOS).

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed as PCOS according to Roterdam (2003) criteria
2. patients with Clomiphene resistance, i.e. failure to ovulate following 100 mg CC for 5 days for at least three cycles.
3. patent fallopian tubes, confirmed by hysterosalpingography or hysteroscopic diagnosis.
4. normal semen analysis parameters of the patients' spouses according to the modified criteria of the World Health Organization.
5. normal serum prolactin, thyroid stimulating hormone and 17-OH progesterone.
6. no systemic disease; no gonadotropin or other hormonal drug treatment during the preceding 3 months.

Exclusion Criteria:

1- Infertility induced by reasons other than PCOS. 2- uterine cavity lesions or ovarian cyst. 3- >40 years old. 4- body mass index (BMI) >26 kg/m2. 5- contraindications to general anesthesia. 6- history of pelvic surgery. 7- other endocrine diseases. 8- a history of liver or kidney disease.

-

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
OVULATION RATE | 7 DAYS BEFORE NEXT MENSES
  SERUM PROGESTERON LEVEL

SECONDARY OUTCOMES:
BIOCHEMICAL PREGNANCY RATE | AFTER 30 DAYS OF INTERVENTION
  BY SERUM HCG
CLINICAL PREGNANCY RATE | AT 6 WEEKS GESTATION
  BY FETAL HEART RATE MONITORING BY ULTRASOUND SCAN

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university maternity hospital, Cairo, Egypt

REFERENCES:
- [Derived] Franik S, Le QK, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for ovulation induction in infertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2022 Sep 27;9(9):CD010287. doi: 10.1002/14651858.CD010287.pub4. PMID 36165742